CLINICAL TRIAL: NCT01231659
Title: Phase II Open Label Study of RAD001 (Everolimus) in Combination With Letrozole in the Treatment of Postmenopausal Women With Locally Advanced or Metastatic, Estrogen Receptor Positive Breast Cancer, After Failure of Tamoxifen and/or Anastrozole and/or Letrozole and/or Fulvestrant and/or Exemestane
Brief Title: Safety and Efficacy of RAD001 (Everolimus) in Combination With Letrozole in the Treatment of Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001JIL05
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Postmenopausal Women; Locally Advanced Metastatic Breast Cancer; Metastatic Breast Cancer
Keywords: RAD001 (Everolimus); Letrozole; Breast cancer; Metastatic Breast cancer; Estrogen receptor positive; Failure of Tamoxifen; Anastrozole or Examestane
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus + Letrozole (Experimental): All patients received 2 tablets (5 mg each) of Everolimus (a total of 10 mg) + 1 tablet of Letrozole (2.5 mg) daily until disease progression or as described in the protocol.
  Interventions: Drug: Everolimus; Drug: Letrozole

INTERVENTIONS:
Drug: Everolimus — Everolimus 10 mg (2 tablets of 5 mg) once daily
  Other Names: RAD001
Drug: Letrozole — Letrozole 2.5 mg once daily

SUMMARY:
This was a multi-center, Israeli phase II open label study evaluating treatment with RAD001 (10 mg daily) combined with letrozole (2.5 mg daily) in postmenopausal women after recurrence or progression on Tamoxifen, Anastrozole or Examestane.

There were no treatments specifically approved after recurrence or progression on AIs. Available options, based on common clinical practice and several treatment guidelines (e.g. NCCN treatment guidelines 2008), included fulvestrant.

Combining RAD001 with letrazole was a rational approach to the treatment of advanced Brest Cancer, offering the potential for inhibition of tumor cell growth\ proliferation and anti angiogenesis while at the same time potentially preventing the development of letrazole resistance.

DETAILED DESCRIPTION:
Screening Period:

Postmenopausal women with estrogen receptor positive, locally advanced or metastatic breast cancer whose disease was refractory to hormonal therapy and had a documented recurrence or progression on last therapy for their breast cancer with either tamoxifen, anastrozole, letrozole, fulvestrant or exemestan were screened for eligibility within 28 days prior to treatment Day 1.

Treatment Period:

Patients started receiving everolimus (10 mg daily oral dose) combined with letrozole (2.5 mg daily oral dose) tablets from treatment Day 1. Study treatment continued until disease progression, intolerable toxicity or consent withdrawal. Dose adjustment (reduction, interruption or possible dose re-escalation to starting dose) could be done based on the safety findings. Tumor assessments were performed every 12 weeks until disease progression. In order to confirm response at least four weeks after first observation, additional scans to determine a complete response (CR) or partial response (PR) or stable disease (SD) were performed. Patients were followed for safety until 28 days after study treatment discontinuation.

Post Treatment Follow up for Survival:

Patients were followed for survival every 3 months for up to 3 years. Survival information could be obtained via phone and information was documented in the source documents.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with estrogen receptor positive locally advanced or metastatic breast cancer after documented recurrence or progression on Tamoxifen, Anastrozole or Examestane.

  * Refractory disease to hormonal therapy is defined as:

    1. Recurrence while on, or within 12 month of end of, adjuvant treatment with Tamoxifen , Anastrozole, or Exemestane.
    2. Recurrence while on, or within 24 month of end of, adjuvant treatment with Letrozole.
    3. Progression while on Tamoxifen, Anastrozole or Exemestane treatment for locally advanced or metastatic breast cancer.

Exclusion Criteria:

* Prior use of chemotherapy and letrozole for Advanced Breast Cancer and mTOR inhibitors as the last anticancer treatment prior to study entry.
* Patients must have radiological evidence of recurrence or progression on last therapy prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-08-09 (Actual); Primary Completion 2012-11-20 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Israel (6):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 7 study centers in Israel.
Pre-assignment Details: Seventy-eight patients were planned to enroll but only 72 patients were actually enrolled and analyzed in this study.
Period: Overall Study
Arm/Group | Everolimus + Letrozole
Started | 72
Per Protocol (PP) Set (All patients that were treated per protocol and analyzed as 1 group) | 72
Safety Set (All patients who received at least 1 dose of the study drug) | 72
Completed | 0
Not Completed | 72
Not completed — Adverse Event | 9
Not completed — Disease Progression | 48
Not completed — Death | 2
Not completed — Patient refused to complete study visit | 1
Not completed — Other protocol defined criteria | 12

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the proportion of patients whose best overall response was either complete response (CR) or partial response (PR) according to RECIST 1.0 for target lesions and assessed by CT: Complete Response (CR), disappearance of all target lesions for a period of at least one month; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (ORR) = CR + PR. Only descriptive statistics.
Time Frame: From the date of randomization until the date of the first documented disease progression or date of death from any cause whichever came first, assessed for approximately 15 months
Population: Per Protocol (PP) Set, which consisted of all patients with measurable disease at baseline, was considered. Only descriptive analysis done.
Measure: Number; unit: Percentage of Participants
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 43
Percentage of Participants | 37.2

2. Secondary Outcome: Median Time to Progression-Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from the date of study entry to the date of first documented tumor progression or death from any cause, whichever occurred first. If a patient did not have an event, PFS was censored at the last date of tumor assessment. For patients with measurable disease at baseline, progression was determined according to the RECIST 1.0 criteria. Only descriptive analysis done.
Time Frame: Date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first, reported between day of first patient randomized up to 66 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Months | 9.0 [0.2 to 59.6]

3. Secondary Outcome: Median Time to Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from the date of study entry to date of death due to any cause. If a death had not observed by the date of analysis, then OS was censored at the date of last contact. Distribution of OS was estimated using the Kaplan Meier method. The median OS along with 95% CI was presented.
Time Frame: From Date of randomization up to approximately 66 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Months | 22.3 [0.2 to 65.0]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was defined as the proportion of patients whose best overall response was either: Complete Response (CR), Partial Response (PR) or Stable Disease (SD). Disease Control Rate was calculated only for patients with measurable disease at baseline and was summarized using descriptive statistics.
Time Frame: From the date of randomization until the date of the first documented disease progression or date of death from any cause whichever came first, assessed for approximately 66 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Percentage of Participants | 85.7 [74.6 to 93.3]

5. Secondary Outcome: Long-term Safety and Tolerability
Description: The assessment of safety was based mainly on the frequency of AEs and on the number of laboratory values that fell outside of pre-determined ranges. Other safety data (e.g. ECG, vital signs) were considered as appropriate. Only descriptive analysis done.
Time Frame: From Date of first dose up to approximately 66 months
Population: Safety Set, which consisted of all patients who received at least 1 dose of the study medication and had at least 1 post-baseline safety evaluation, was considered. Only descriptive analysis done.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Participants
  AEs - All | 72
  AEs - Grade 3 | 39
  AEs - Grade 4 | 7

6. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 2002 days (treatment duration ranged from 1 to 1974 days).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 2092 days. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 2002 days (on-treatment), up to approximately 2092 days (study duration)
Population: Clinical database population (all treated patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Letrozole
Number analyzed (Participants) | 72
Participants
  On-treatment deaths | 2
  Post-treatment deaths | 50
  All deaths | 52

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from First Patient First Treatment (FPFT) up to 28 days after study drug discontinuation, for a maximum duration of 2002 days (treatment duration ranged from 1 to 1974 days).
Description: Any sign or symptom that occurs during the study treatment and 28 days post treatment follow up.
Arm/Group | Everolimus + Letrozole
All-Cause Mortality (participants affected / at risk) | 2/72
Serious Adverse Events (participants affected / at risk) | 26/72
Other Adverse Events (participants affected / at risk) | 71/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Letrozole (N=72)
Anaemia (Blood and lymphatic system disorders) | 5
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Hypercalcaemia (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Death (General disorders) | 1
Disease progression (General disorders) | 2
Infusion related reaction (General disorders) | 1
Pyrexia (General disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Angiodysplasia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Letrozole (N=72)
Anaemia (Blood and lymphatic system disorders) | 21
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 21
Dry mouth (Gastrointestinal disorders) | 9
Gingival pain (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 15
Oral pain (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 27
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 5
Chest pain (General disorders) | 4
Disease progression (General disorders) | 16
Fatigue (General disorders) | 49
Influenza like illness (General disorders) | 18
Local swelling (General disorders) | 4
Mucosal inflammation (General disorders) | 23
Oedema peripheral (General disorders) | 18
Pyrexia (General disorders) | 16
Pharyngitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 11
Viral infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 10
Blood creatinine increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 8
Weight decreased (Investigations) | 21
White blood cell count decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 19
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 15
Headache (Nervous system disorders) | 22
Insomnia (Psychiatric disorders) | 8
Pelvic pain (Reproductive system and breast disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 8
Nail ridging (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 22
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 8
Lymphoedema (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.